CLINICAL TRIAL: NCT07036796
Title: Effect of Melatonin on the Clinical Outcomes in Type 2 Diabetic Patients With Peripheral Neuropathy
Brief Title: Effect of Melatonin in Patients With Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, manar magdy, Demonstrator at Ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC#310
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetic Neuropathy; Diabetic Peripheral Neuropathy in Type 2 Diabetic Patients
Keywords: Diabetic peripheral neuropathy; Diabetic neuropathies; Diabetic neuropathy in type 2 diabetes; Melatonin
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Prospective Randomized controlled clinical trial open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Melatonin group (Active Comparator): Group 1: Melatonin group (n=30) Patients will receive 10 mg (2 5mg Capsules) 1 hour before bedtime for 12 weeks, in addition to the standard therapy.
  Interventions: Drug: Melatonin
- Group 2: control group (No Intervention): Group 2: No intervention, (n=30) patients will receive only standard therapy for 12 weeks

INTERVENTIONS:
Drug: Melatonin — Melatonin (N-acetyl-5-methoxytryptamine), also called the hormone of darkness, secreted primarily by the pineal gland. Possesses antioxidant, anti-inflammatory, anti-diabetic and neuroprotective effects. All of which could be explained by its activation of Nrf2 signaling pathway.
  Melatonin administration has shown to improve motor nerve conduction velocity and nerve blood flow, reduce the levels of pro-inflammatory cytokines, reinforce antioxidant defense, and decrease DNA fragmentation through upregulating nrf2 pathway, when tested in mice with diabetic peripheral neuropathy. Moreover, early treatment with melatonin has shown to prevent developing diabetic neuropathy in streptozotocin induced diabetic mice.
  Arms: Group 1: Melatonin group

SUMMARY:
The aim of the current study is to measure the effect of melatonin as adjunct therapy on oxidative stress, inflammatory markers and clinical outcome in type 2 diabetic patients with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Diabetic neuropathy is a microvascular complication affecting 50% of patients throughout their lifetime. It leads to various complications including foot ulcerations and lower limb amputations, thus impairs the patient's quality of life. Distal symmetrical polyneuropathy is the most common subtype. Symptoms include tingling, burning and electrical pain associated with nocturnal exacerbation. Almost 50% of patients are asymptomatic thus diagnosis must include assessment of signs.

Pathophysiologic mechanism behind hyperglycemia induced nerve damage include the activation of various pathways including polyol and advanced glycation end product (AGE), which produces reactive oxygen species. Molecular studies have revealed the involvement of certain transcriptional regulators such as Nrf2-Keap1 and NfKb inflammatory cascade.

Nuclear erythroid growth factor-2 (Nrf2) functions primarily as a defense mechanism in cellular oxidative stress, producing anti-oxidant enzymes as glutathione reductase (GSH) and superoxide dismutase (SOD). However, in long term hyperglycemia, downregulation of nrf2 takes place, leading to accumulation of reactive oxygen species (ROS), which in turn activates nfkb inflammatory pathway and produces various cytokines such as tumor necrosis factor-alpha (Tnf-alpha), interleukin-1 (IL-1) and interleukin-6 (IL-6). Tumor-necrosis factor is known to be highly associated with nerve damage.

Drugs that target disease pathophysiology are currently unavailable, instead DPN management mainly depends on lifestyle modification through weight loss, blood pressure, blood glucose, lipid profile management along with symptomatic care. Yet these fail to stop disease progression.

Melatonin is known to possess anti-oxidant and anti-inflammatory properties through upregulating nrf2. It's hypothesized that adding it to standard therapy shall activate nrf2, and downregulate nfkb pathway and inflammatory cytokines, improving disease progression and patient's quality of life.

The aim of the current study is to measure the effect of melatonin on oxidative stress, inflammatory markers and clinical outcome in type 2 diabetic patients with DPN.

All patients will be assessed for the following data at baseline:

1. Age, gender, diabetes duration, diabetic neuropathy duration.
2. HbA1c, liver functions, kidney functions and lipid profile.

Lab assessment will be done at both baseline and at the end of the trial to assess the effect of melatonin on the following:

1. Nuclear erythroid related factor-2 (NRf2) (an oxidative marker)
2. Tumor necrosis factor-alpha (an inflammatory marker)

Assessment of clinical outcomes will be done as well, at both baseline and endpoint using the following:

1. Toronto clinical scoring system (TCSS)
2. Michigan neuropathy screening instrument questionnaire (MNSIQ) Samples used to assess oxidative and inflammatory markers will be stored at -80 degrees to be analyzed later at the end of the study using ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 40-75 years diagnosed with type 2 DM.
2. Diabetes duration at least 1 year.
3. Patients diagnosed with diabetic peripheral neuropathy.
4. Stable antidiabetic medication for at least 1 month before enrollment and during the trial

Exclusion Criteria:

1. Patients with autoimmune disorders (such as lupus and rheumatoid arthritis), thyroid diseases, peripheral arterial disease and cancer patients.
2. Patients with severe kidney or liver dysfunction.
3. Patients diagnosed with neurodegenerative diseases.
4. Active infection.
5. Use of medications or supplements known to cause or treat peripheral neuropathy.
6. Alcohol consumption or substance abuse.
7. Patients consuming any antioxidant supplements or anti-inflammatory medicines during or 3 months before enrollment.
8. Pregnancy or lactation or expecting to get pregnant during the study.
9. Allergy to melatonin.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-07-04 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
Concentration of human nuclear factor erythroid 2-related factor (Nrf2) | Change from baseline human Nuclear factor erythroid 2-related factor at 3 months.
  Oxidative stress marker

SECONDARY OUTCOMES:
Concentration of Tumor necrosis factor alpha | Change from baseline Tumor necrosis factor alpha at 3 months
  Inflammatory marker
Michigan neuropathy screening instrument questionnaire (MNSI-Q) | At baseline and after 3 months
  A questionnaire of 15 yes or no questions, a score of 7 or more means more neuropathic symptoms
Toronto clinical scoring system (TCSS) | At baseline and after 3 months
  A scoring system used to assess symptoms, reflexes and signs, as score increases indicates more neuropathy.
Diabetic neuropathy score (DNS) | At baseline and after 3 months
  A score used to assess the major symptoms of DPN.
D-39 questionnaire | At baseline and after 3 months.
  A questionnaire used to test the effect of diabetes on patient's quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided